CLINICAL TRIAL: NCT04614610
Title: Randomized Trial Evaluating Lidocaine Intravenous in the Emergency Department For Sickle Cell Crisis - RELIEF-SCC
Brief Title: Lidocaine Intravenous in the Emergency Department For Sickle Cell Crisis
Acronym: RELIEF-SCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Community Medical Center, Toms River, NJ (Other)
Collaborators: Newark Beth Israel Medical Center (Other); Monmouth Medical Center (Other); Rutgers Robert Wood Johnson Medical School (Other)
Responsible Party: Principal Investigator, Andrew Vassallo, Primary Research Coordinator, Community Medical Center, Toms River, NJ
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-58
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell Disease; Sickle Cell Crisis; Pain, Acute
Keywords: lidocaine; ALTO; sickle cell pain
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Acute Pain

STUDY DESIGN:
Intervention Model Description: Patients presenting to the emergency department for an acute sickle cell crisis who are refractory to one dose of intravenous opiate therapy will be randomized to either lidocaine 1.5mg/kg (max: 200mg) or matching dextrose placebo along with either morphine 0.1-0.15mg/kg IV or hydromorphone 0.01-0.02mg/kg IV.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Lidocaine or placebo will be dispensed from the pharmacy in identical bags labeled "Lidocaine (x)mg or Placebo". The pharmacy will maintain randomization and blinding until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine 1.5mg/kg (Max: 200mg) in dextrose 5% 100mL over 10 minutes along with either morphine 0.1-0.15mg/kg IV OR hydromorphone 0.01-0.02mg/kg IV.
  Interventions: Drug: Lidocaine Iv
- Placebo (Placebo Comparator): Dextrose 5% 100mL (placebo) over 10 minutes along with either morphine 0.1-0.15mg/kg IV OR hydromorphone 0.01-0.02mg/kg IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Iv — Lidocaine 1.5mg/kg (Max dose: 200mg) in Dextrose 5% 100mL over 10 minutes
  Arms: Lidocaine
Drug: Placebo — Dextrose 5% 100mL over 10 minutes
  Arms: Placebo

SUMMARY:
Sickle cell crisis continues to be a frequent presentation to emergency departments. Patients presenting will often require immediate treatment for their pain and often times this will include opioids. The opioid epidemic has cost thousands of lives; and continues to be a significant problem posing several challenges when treating patients presenting with sickle cell disease. Primarily, opioids remain the mainstay of treatment for these patients and the push to address the opioid crisis may present challenges for adequate opioid administration in patients suffering from a sickle cell crisis while hospitals find ways to curb the opioid crisis overall. Opioid treatment for patients in acute vaso-occlusive crisis has significantly contributed to quality of life and life expectancy of patients with this diagnosis. Measures should continue to attempt to administer a multi-model approach to sickle cell patients to minimize the morphine milligram equivalents in these patients while also successfully addressing the patient's pain. IV lidocaine is a pain medication that has been evaluated in several painful experiences, such as in renal colic. A few case reports have shown IV lidocaine use in sickle cell can be a potential effective adjunct medication to opioids to treat pain and reduce further opioid requirements. Currently, no prospective controlled trial exists to evaluate the true benefit of IV lidocaine in this population. Our study aims to evaluate IV lidocaine as an adjunct to opioid treatment in the emergency department to determine if improved pain is achieved and if there is a reduction in overall morphine milligram equivalents throughout the emergency department visit.

DETAILED DESCRIPTION:
Pain is the most frequent reason for emergency department visits in the United States, especially for those patients with sickle cell disease (SCD). Painful vaso-occlusive events frequently require admission to the hospital despite opioid therapy, which is the mainstay of treatment for moderate to severe pain in SCD. Achieving adequate pain control with escalating doses of opioid analgesics may be difficult due to tolerance, physical dependence, and side effects. Common side effects include pruritus, nausea and vomiting, constipation, urinary retention, sedation, and respiratory depression. With the recent focus on the opiate crisis there has been a push towards the use of alternative to opiates (ALTO) for a variety of pain syndromes.

Lidocaine is a class 1b sodium channel blocking agent that is typically used as an anti-arrhythmic and local anesthetic. This medication also has potent anti-inflammatory, anti-hyperalgesic, and gastrointestinal pro-peristaltic properties. Lidocaine may be useful as an adjunct to opioids in response to a painful sickle cell crisis. Intravenous (IV) lidocaine infusion has previously shown benefit in neuropathic pain, renal colic, and peri-operative pain. No prospective studies have evaluated lidocaine for SCD pain thus far.

A previous retrospective study evaluated lidocaine infusion as adjuvant therapy to patients with SCD. Eleven patients were given a total of 15 IV lidocaine trials. Investigators found clinical improvement in pain score from pre-lidocaine challenge to 24 hours post (defined as a >20% reduction in pain scores) in 53.3% (8 of 15) of patients. Of the 8 clinically successful trials, the mean reduction in morphine dose equivalents (MDE) from 24 hours pre to 24 hours post lidocaine was 32.2%. Two patients experienced disorientation and dizziness. The authors concluded that lidocaine was able to provide pain relief and reduce the amount of morphine necessary during SCD vaso-occlusive crisis and that prospective studies are needed to determine its true efficacy, dosing, and tolerability.

A prospective, single-arm, phase II trial evaluated lidocaine 5% patches for neuropathic pain and pain related to vaso-occlusive sickle cell crises in children ages 6 to 21 years old. Patches were applied to the painful area for 12 hours a day. The primary endpoint was the proportion of inpatients with significant pain relief defined as a decrease of at least 2 points on the visual analog pain scale (VAS, from 0-10) measured at 12 hours after patch placement over two consecutive days. The use of additional treatments such as antiepileptics and opioids were allowed and their usage was documented. The primary outcome of VAS improvement of >2 over 2 consecutive days was observed in 48.6% of evaluated patients (19/39). Transdermal lidocaine was tolerated well with only 3 minor adverse events reported (two localized skin reactions and one generalized skin eruption) and no serious adverse events.

The theoretical benefits along with the two previously discussed studies provide evidence to further investigate the use of lidocaine in SCD pain. Studies are needed to know whether lidocaine may be able to benefit alleviate pain quicker and minimize need for opiates similarly to its use in renal colic. This prospective trial aims to evaluate whether lidocaine can decrease the opiate needs during a SCD crisis while providing adequate pain relief and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old with sickle cell disease experiencing persistent severe (7-10/10) pain despite receiving at least one dose of intravenous opiate analgesic.

Exclusion Criteria:

* Patients < 18 years old and pregnant
* Patients presenting with or suspected to have acute chest syndrome
* Allergy or intolerance to lidocaine products or morphine/hydromorphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain at 30 minutes | from pre-lidocaine infusion to 30 minutes post-infusion
  Change of visual analog pain scale (VAS, 0-10) at 30 minutes post-infusion of lidocaine or placebo.

SECONDARY OUTCOMES:
Total opiate dosage received | from presentation to the Emergency department (ED) until patient disposition (up to 12 hours)
  Total morphine mg equivalents (MME) of opiate received normalized to patient's bodyweight during their ED stay.
% Patients requiring additional opiate administration | from presentation to the Emergency department (ED) until patient disposition (up to 12 hours)
  Percentage of patients requiring an additional opiate after the lidocaine vs. placebo.
Time to next opiate administered | from administration of lidocaine infusion until patient disposition (up to 12 hours) or next opiate administered
  Time (minutes) until next opiate is administered after lidocaine vs. placebo.
Total MME post-lidocaine up to 12 hours | 12 hours post-lidocaine or placebo infusion.
  Total MME needed after lidocaine vs placebo up to 12 hours
Percentage of patients discharged from ED | from presentation to the Emergency department (ED) until patient disposition (up to 12 hours)
  Percentage of patients discharged from the ED.
Percentage of patients receiving a >20% reduction in pain scale | from presentation to the Emergency department (ED) until patient disposition (up to 12 hours)
  Percentage of patients receiving a >20% reduction in pain scale based on the VAS (0-10).
Change in visual analog pain scale (VAS, 0-10 with 10 being the most pain) at 60 and 90 minutes | 60 and 90 minutes
  Change in VAS at 60 and 90 minutes post-infusion.
Number of adverse effects of treatment | from presentation to the Emergency department (ED) until patient disposition (up to 12 hours)
  Reported adverse effects during study treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Shreni Zinzuwadia, MD, Principal Investigator — Newark Beth Israel
Locations (3):
- United States (3):
  - Monmouth Medical Center, Long Branch, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] E Silva LOJ, Scherber K, Cabrera D, Motov S, Erwin PJ, West CP, Murad MH, Bellolio MF. Safety and Efficacy of Intravenous Lidocaine for Pain Management in the Emergency Department: A Systematic Review. Ann Emerg Med. 2018 Aug;72(2):135-144.e3. doi: 10.1016/j.annemergmed.2017.12.014. Epub 2018 Feb 1. PMID 29395284
- [Background] Lanzkron S, Carroll CP, Haywood C Jr. The burden of emergency department use for sickle-cell disease: an analysis of the national emergency department sample database. Am J Hematol. 2010 Oct;85(10):797-9. doi: 10.1002/ajh.21807. PMID 20730795
- [Background] Payne J, Aban I, Hilliard LM, Madison J, Bemrich-Stolz C, Howard TH, Brandow A, Waite E, Lebensburger JD. Impact of early analgesia on hospitalization outcomes for sickle cell pain crisis. Pediatr Blood Cancer. 2018 Dec;65(12):e27420. doi: 10.1002/pbc.27420. Epub 2018 Aug 27. PMID 30151977
- [Background] Lexicomp Online, Lexi-Drugs Online, Hudson, Ohio: Lexi-Comp, Inc.; December 15, 2017.
- [Background] Eipe N, Gupta S, Penning J. Intravenous Lidocaine for Acute Pain: an Evidence-based Clinical Update. BJA Education,16(9):292-298(2016). Doi: 10.1093/bjaed/mkw008
- [Background] Carroll CP, Lanzkron S, Haywood C Jr, Kiley K, Pejsa M, Moscou-Jackson G, Haythornthwaite JA, Campbell CM. Chronic Opioid Therapy and Central Sensitization in Sickle Cell Disease. Am J Prev Med. 2016 Jul;51(1 Suppl 1):S69-77. doi: 10.1016/j.amepre.2016.02.012. PMID 27320469
- [Background] Nguyen NL, Kome AM, Lowe DK, Coyne P, Hawks KG. Intravenous Lidocaine as an Adjuvant for Pain Associated with Sickle Cell Disease. J Pain Palliat Care Pharmacother. 2015;29(4):359-64. doi: 10.3109/15360288.2015.1082009. PMID 26654408
- [Background] Rousseau V, Morelle M, Arriuberge C, Darnis S, Chabaud S, Launay V, Thouvenin S, Roumenoff-Turcant F, Metzger S, Tourniaire B, Marec-Berard P. Efficacy and Tolerance of Lidocaine 5% Patches in Neuropathic Pain and Pain Related to Vaso-occlusive Sickle Cell Crises in Children: A Prospective Multicenter Clinical Study. Pain Pract. 2018 Jul;18(6):788-797. doi: 10.1111/papr.12674. Epub 2018 Feb 28. PMID 29266772
- [Background] Soleimanpour H, Hassanzadeh K, Vaezi H, Golzari SE, Esfanjani RM, Soleimanpour M. Effectiveness of intravenous lidocaine versus intravenous morphine for patients with renal colic in the emergency department. BMC Urol. 2012 May 4;12:13. doi: 10.1186/1471-2490-12-13. PMID 22559856
- [Background] Firouzian A, Alipour A, Rashidian Dezfouli H, Zamani Kiasari A, Gholipour Baradari A, Emami Zeydi A, Amini Ahidashti H, Montazami M, Hosseininejad SM, Yazdani Kochuei F. Does lidocaine as an adjuvant to morphine improve pain relief in patients presenting to the ED with acute renal colic? A double-blind, randomized controlled trial. Am J Emerg Med. 2016 Mar;34(3):443-8. doi: 10.1016/j.ajem.2015.11.062. Epub 2015 Dec 1. PMID 26704774
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Holdgate A, Asha S, Craig J, Thompson J. Comparison of a verbal numeric rating scale with the visual analogue scale for the measurement of acute pain. Emerg Med (Fremantle). 2003 Oct-Dec;15(5-6):441-6. doi: 10.1046/j.1442-2026.2003.00499.x. PMID 14992058
- [Background] Motov S, Fassassi C, Drapkin J, Butt M, Hossain R, Likourezos A, Monfort R, Brady J, Rothberger N, Mann SS, Flom P, Gulati V, Marshall J. Comparison of intravenous lidocaine/ketorolac combination to either analgesic alone for suspected renal colic pain in the ED. Am J Emerg Med. 2020 Feb;38(2):165-172. doi: 10.1016/j.ajem.2019.01.048. Epub 2019 Jan 30. PMID 30770244